CLINICAL TRIAL: NCT03091361
Title: A Prospective, Single-blind Evaluation of the Positive Predictive Value (PPV) of the MolecuLight i:X™ Imaging Device to Predict the Presence of Bacteria in Chronic Wounds
Brief Title: Post Market Clinical Followup of MolecuLight i:X's PPV to Predict Presence of Bacteria in Wounds
Status: Completed | Type: Observational
Sponsor: MolecuLight Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-101
Record Dates: First submitted 2016-11-08; First posted 2017-03-27 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Wounds and Injuries
Keywords: Bacterial imaging; PPV; Chronic wounds
MeSH Terms: conditions — Wounds and Injuries | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients (imaging/no intervention): There is only one group in this study, the imaging/no intervention group. These patients will meet all enrollment criteria and bacterial (red or cyan) fluorescence will be visualized within or around their wound with the MolecuLight i:X imaging device. A targeted curettage sample will be taken from the site of fluorescence and sent for microbiological analysis. There will be no intervention or followup.
  Interventions: Other: imaging, no intervention

INTERVENTIONS:
Other: imaging, no intervention — no intervention

SUMMARY:
This is a non-randomized, single-blind post market clinical follow-up study for which 50 patients will be imaged at the Judy Dan Research and Treatment Centre who present with a chronic and are receiving standard wound care treatment. The i:X imaging device visualizes fluorescing bacteria in real-time. The device will be used as an adjunctive tool in the assessment of the wound and will be used to guide the targeted sampling of a wound (with curettage scraping). The overall objective of this work is to evaluate the positive predictive value (PPV) of the MolecuLight i:X Imaging Device in predicting the presence of bacteria in chronic wounds. The presence of bacteria will be determined micro-biologically by semi-quantitative culture analysis.

DETAILED DESCRIPTION:
MolecuLight Inc. (Toronto, Canada) has recently introduced to the Canadian market an innovative imaging device, the MolecuLight i:X™ Imaging Device, that offers real-time detection of important biological and molecular information of a chronic wound, and could have significant impact on improving conventional wound care and management. The MolecuLight i:X Imaging Device is intended to assist clinicians during care and management of patients with chronic wounds by screening for the presence of potentially harmful bacteria levels. The device can capture and document either an image or video of the chronic wound where the presence of fluorescent bacteria appears under violet light illumination. This information can be used to guide a clinician to inspect, sample, debride or further evaluate areas within or around a wound where fluorescent bacteria are present. Though the MolecuLight i:X Imaging Device has been shown to be effective in controlled settings, this study is deploying the device in a larger population and evaluating the ability of the MolecuLight i:X device to positively predict the presence of bacteria in chronic wounds.

The overall objective of this work is to evaluate the MolecuLight i:X Imaging Device in screening of chronic wounds for the presence of bacteria. The device is intended to guide the clinician to inspect, sample, debride or further evaluate areas within or around a wound where fluorescent bacteria are present.

All imaging will be performed with the MolecuLight i:X Imaging Device at an appropriate distance from the wound of interest (8 - 12 cm), which is indicated by the range finder LED. Illumination is provided by two violet (405 nm) LEDs that produce a bright, but clinically safe, uniform illumination. Fluorescence imaging is performed on the camera in real-time while the device is in fluorescence mode and the room lights are turned off. If room ambient light cannot be eliminated to an acceptable level (indicated by the ambient light sensor), the MolecuLight drape must be used to achieve a dark environment. A standard measurement sticker will be placed adjacent to the wound within the field of view to act as a reference for size.

All microbiological analysis will be performed as per clinic standard practice. Tissue samples will be analyzed for culture and sensitivity, yielding the species of bacteria present in the sample (if any), the susceptibility to various antibiotics and a measure of the bacterial load.

ELIGIBILITY:
Inclusion Criteria:

* presents with a chronic wound of the lower limb (e.g. diabetic foot ulcer, venous leg ulcer, other acceptable aetiology)
* red or cyan fluorescence signals observed within or around wound on MolecuLight i:X images

Exclusion Criteria:

* Treatment with an investigational drug within 1 month before study enrollment
* Use of systemic (oral or intravenous) antibiotics
* Inability to consent to medical photography
* Any contra-indication to routine wound care and/or monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving routine wound care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Linden, MD, Principal Investigator — Judy Dan Research and Treatment Center
Locations (1):
- Judy Dan Research and Treatment Centre, North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rennie MY, Lindvere-Teene L, Tapang K, Linden R. Point-of-care fluorescence imaging predicts the presence of pathogenic bacteria in wounds: a clinical study. J Wound Care. 2017 Aug 2;26(8):452-460. doi: 10.12968/jowc.2017.26.8.452. PMID 28795890

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients (Imaging/no Intervention)
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients (Imaging/no Intervention)
Number analyzed (Participants) | 30
Age, Customized [Count of Participants; unit: Participants] | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Region of Enrollment [Number; unit: participants]
  Canada | 30

OUTCOME MEASURES:

1. Primary Outcome: Positive Predictive Value (PPV) of Localized Red Fluorescence Signals With Microbiological Samples
Description: PPV reflects the probability that a region of red fluorescence within or around a wound will contain bacteria. Meaning the number cases where qPCR analysis of wound tissue biopsies from red fluorescent region showed to have pathogen load ≥ 104 CFU/g divided by the total number of cases where red florescence was observed in the wound multiplied by 100,
Time Frame: 3 months
Measure: Number; unit: percentage of PPV of red fluorescence
Arm/Group | All Patients (Imaging/no Intervention)
Number analyzed (Participants) | 30
percentage of PPV of red fluorescence | 100

ADVERSE EVENTS:
Arm/Group | All Patients (Imaging/no Intervention)
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No